CLINICAL TRIAL: NCT00946322
Title: Couple-Based Treatment for Alcohol Use Disorders and PTSD
Brief Title: Couple-Based Treatment for Alcohol Use Disorders and Post-Traumatic Stress Disorder
Acronym: CTAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDA-2-019-09S
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Alcohol-related Disorders; Post-traumatic Stress Disorder
Keywords: post-traumatic stress disorder; alcohol-related disorders; substance use disorders; couple therapy
MeSH Terms: conditions — Alcohol-Related Disorders; Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: CTAP (Experimental): Couple-Based Treatment for Alcohol Use Disorders and PTSD
  Interventions: Behavioral: Couple-Based Treatment for Alcohol Use Disorders and PTSD

INTERVENTIONS:
Behavioral: Couple-Based Treatment for Alcohol Use Disorders and PTSD — This intervention includes cognitive-behavioral strategies for helping couples to reduce alcohol use and PTSD, while improving relationship functioning.
  Other Names: CTAP

SUMMARY:
The purpose of this study is to develop and test a couple-based treatment for Veterans with an alcohol use disorder and post-traumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* Veteran must meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV; American Psychiatric Association, 1994) criteria for current (past 12 months) alcohol abuse or dependence and alcohol must be the Veteran's primary substance of abuse as determined by a clinical algorithm (Fals-Stewart, Stappenbeck et al, 2004);
* Veteran must meet DSM-IV criteria for current (past month) PTSD;
* Veteran consumed alcohol in the past 90 days;
* couple must be married to or living with their current partner for at least 1 year;
* Veteran agrees to a goal of abstinence from drugs at least for the duration of the 15-week study-based treatment;
* Veteran agrees to the goal of abstaining from alcohol or consuming alcohol within low risk drinking guidelines during the duration of the 15-week study-based counseling;
* Veteran agrees to forego other treatment for alcohol-related disorders except for self help meetings (e.g., AA) or treatment required for a clinical emergency or clinical deterioration for the duration of the 15-week study based treatment;
* Veteran agrees to forgo other PTSD treatment except for treatment required for a clinical emergency or clinical deterioration for the duration of the 15-week study based treatment;
* couple agrees to forgo other couple-based counseling for the duration of the 15-week study based treatment except for treatment required for a clinical emergency or clinical deterioration;
* partner does not meet DSM-IV criteria for current (past 12 month) substance use disorder (other than nicotine)
* partner does not meet DSM-IV criteria for current (past month) PTSD.

Exclusion Criteria:

* Veteran has dependence on alcohol or other drugs that requires inpatient treatment or medical detoxification (as indicated by daily heavy use or use to prevent or deal with withdrawal symptoms) - after completing detoxification, Veteran may be eligible for the study;
* Veteran or partner are at immediate risk for suicide or homicide (current plan or intent);
* Veteran or partner exhibit a history of suicide or homicide attempt in the past year;
* Veteran is participating in a methadone maintenance or suboxone maintenance program and is seeking treatment for adjunctive outpatient services;
* Veteran or partner meets DSM-IV criteria for a current organic mental disorder, schizophrenia, delusional (paranoid) disorder, or any of the other psychotic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah A. Schumm, PhD, Principal Investigator — Cincinnati VA Medical Center, Cincinnati, OH
Locations (1):
- Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 couple was excluded due to discovery that they did not meet eligibility requirements
Period: Pre-treatment
Arm/Group | Arm 1: CTAP
Started | 12
Completed | 11
Not Completed | 1
Not completed — participant failure to follow up | 1
Period: Post-treatment
Arm/Group | Arm 1: CTAP
Started | 11
Completed | 9
Not Completed | 2
Not completed — participant failure to follow up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.22 (16.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Clinician-administered PTSD Scale (CAPS)
Description: Total severity score on the CAPS was used. Higher = worse outcome. Possible range of scores 0-135.
Time Frame: Pre- to post-treatment (~20 weeks)
Population: Participants completing both pre- and post-treatment assessments were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 9
units on a scale
  Pre-treatment | 58.89 (17.57)
  Post-treatment | 40.22 (24.30)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-test; Test type: Superiority or Other; p = .028, t-test, 2 sided

2. Primary Outcome: Percentage Days of Heavy Drinking
Description: Percentage days of heavy drinking (PDHD) was calculated by dividing the number of days in which the Veteran consumed more than six standard drinks by the total days in the period. Both partners reported upon the Veterans' drinking behaviors. Following common practice in AUD research (e.g., McCrady, Epstein, Cook, Jensen, & Hildebrandt, 2011), we used the highest report of the two regarding PDHD to reduce possible underreporting. Possible range of scores 0-100%. Higher = worse.
Time Frame: Pre- to post-treatment (~20 weeks)
Population: Participants completing pre- and post-treatment assessments were analyzed
Measure: Mean (Standard Deviation); unit: percentage of days of heavy drinking
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 9
percentage of days of heavy drinking
  Pre-treatment | 29.01 (39.16)
  Post-treatment | 16.19 (29.74)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-tests were used. Due to variable skewness, variables were logarithm-transformed to improve their distributions; Test type: Superiority or Other; p = .022, t-test, 2 sided

3. Secondary Outcome: Patient-reported Beck Depression Inventory - II (BDI-II)
Description: Patient-reported total severity score on Beck Depression Inventory - II (BDI-II). Possible range 0-63. Higher = worse.
Time Frame: Pre- to post-treatment
Population: Participants completing the BDI-II at pre- and post-treatment were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 7
units on a scale
  Pre-treatment | 27.81 (13.89)
  Post-treatment | 17.62 (15.18)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-test; Test type: Superiority or Other; p = .043, t-test, 2 sided

4. Secondary Outcome: Patient-reported Dyadic Adjustment Scale
Description: Patient-reported total score on the Dyadic Adjustment Scale (DAS), which is a measure of couple relationship satisfaction. Possible range = 0 - 151. Higher = worse.
Time Frame: Pre- to post-treatment (~20 weeks)
Population: Participants completing pre- and post-treatment assessment were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 9
units on a scale
  Pre-treatment | 96.12 (25.04)
  Post-treatment | 100.76 (24.10)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-test; Test type: Superiority or Other; p = .482, t-test, 2 sided

5. Primary Outcome: Patient-reported PTSD Checklist
Description: Patient self-reported total severity score on the PTSD Checklist - Specific (PCL-S) version. Possible range of scores 17-85. Higher = worse.
Time Frame: Pre- to post-treatment (~20 weeks)
Population: Participants completing pre- and post-treatment assessments were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 9
units on a scale
  Pre-treatment | 57.72 (13.18)
  Post-treatment | 43.78 (17.26)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-test; Test type: Superiority or Other; p = .009, t-test, 2 sided

6. Primary Outcome: Partner-reported PTSD Checklist
Description: Partner-reported total severity score for patient's PTSD symptoms on the PTSD Checklist - Specific (PCL-S) version. Possible range 17-85. Higher = worse.
Time Frame: Pre- to post-treatment (~20 weeks)
Population: Participants completing pre- and post-treatment assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 9
units on a scale
  Pre-treatment | 54.89 (14.31)
  Post-treatment | 35.67 (14.67)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-test; Test type: Superiority or Other; p = .001, t-test, 2 sided

7. Secondary Outcome: Partner-reported Beck Depression Inventory - II
Description: Partner-reported Beck Depression Inventory - II (BDI-II) total severity score. Possible range 0-63. Higher = worse.
Time Frame: Pre- to post-treatment (~20 weeks)
Population: Participants completing the pre- and post-treatment assessment were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 7
units on a scale
  Pre-treatment | 12.63 (9.15)
  Post-treatment | 6.41 (9.87)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-test; Test type: Superiority or Other; p = .027, t-test, 2 sided

8. Secondary Outcome: Partner-reported Dyadic Adjustment Scale
Description: Partner-reported total score on the Dyadic Adjustment Scale, which is a measure of couple relationship satisfaction. Possible range 0-151. Higher = worse.
Time Frame: Pre- to post-treatment (~20 weeks)
Population: Participants completing pre- and post-treatment assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: CTAP
Number analyzed (Participants) | 9
units on a scale
  Pre-treatment | 92.85 (30.08)
  Post-treatment | 101.49 (21.54)
Statistical Analysis 1: Comparison: Arm 1: CTAP; Paired sample t-test; Test type: Superiority or Other; p = .177, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During duration of treatment and through post-treatment assessment (~20 weeks)
Arm/Group | Arm 1: CTAP
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Study was an initial open-trial pilot study. A causal relationship cannot be determined between study interventions and outcomes due to lack of a comparison condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes